CLINICAL TRIAL: NCT02995369
Title: DryShield vs Cotton Roll Isolation During Sealants Placement: Efficiency and Patient
Brief Title: DryShield vs Cotton Roll Isolation During Sealants Placement: Efficiency and Patient Preference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Nuntiya Kakanantadilok, Director Division of Pediatric Dentistry, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-7229
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-11

CONDITIONS: Time; Patient Preference
Keywords: Sealants; Dryshield; Cotton roll; Isolation; Efficiency; Preference
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cotton Roll Isolation (left), then DryShield Isolation (right) (Experimental): Cotton rolls (CRI) will be used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using Dryshield (DS) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second).
  Interventions: Device: DryShield; Other: Cotton rolls
- Cotton Roll Isolation (right), then DryShield Isolation (left) (Experimental): Cotton rolls (CRI) will be used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using DryShield (DS) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second).
  Interventions: Device: DryShield; Other: Cotton rolls
- DryShield Isolation (left), then Cotton Roll Isolation (right) (Experimental): DryShield (DS) will be used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second).
  Interventions: Device: DryShield; Other: Cotton rolls
- DryShield Isolation (right), then Cotton Roll Isolation (left) (Experimental): DryShield (DS) will be used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second).
  Interventions: Device: DryShield; Other: Cotton rolls

INTERVENTIONS:
Device: DryShield — DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
Other: Cotton rolls — Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water is used.

SUMMARY:
The goals of this study are to determine if 1) placement times of pit and fissure sealants using the DryShield system differ from those when using the cotton roll isolation technique; and 2) there is a significant difference in patient preference between Dryshield and the cotton roll technique.

DETAILED DESCRIPTION:
Pit and fissure caries account for 80 to 90 percent of all caries in permanent posterior teeth. Pit-and-fissure sealants can be used effectively to prevent caries. By micromechanically bonding to the teeth, they provide a physical barrier that keeps microorganisms and food particles from collecting in susceptible pits and fissures, thus preventing caries initiation and arresting caries progression. The effectiveness of sealants for caries prevention depends on long-term retention, which is largely a function of meticulousness of application: keeping the tooth surface free from saliva contamination during application and polymerization is critical. Low retention of sealants has been attributed to insufficient moisture control. Therefore, proper isolation of the teeth is one of the most important steps when placing sealants to ensure their retention. Cotton roll isolation (CRI) has been widely used for sealant placement, and is the most common method among pediatric dentists. Although very effective, CRI can be a challenging technique especially when used in young children: the cotton rolls can be cumbersome for both the patient and the clinician. A previous study demonstrated that new moisture control systems such as Isolite, produce sealant retention rates comparable to cotton roll isolation, while decreasing procedure time. DryShield (DS) has recently been introduced as an all-in-one isolation system. It is similar to the Isolite as it combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block, but differs in that it's autoclavable and does not provide illumination. Its design allows it to suction and isolate half the oral cavity at a time. Therefore, it should presumably facilitate sealants placement under a more controlled environment, while reducing chair time for the dentist.

The goals of this study are to determine if 1) placement times of pit and fissure sealants using the DryShield system differ from those when using the cotton roll isolation technique; and 2) there is a significant difference in patient preference between DryShield and the cotton roll technique.

ELIGIBILITY:
The target population will include healthy, cognitively normal patients who present to one of the Montefiore pediatric dental clinics for an intake or a recall visit who are determined to benefit from sealants application, or patients who present solely for a sealant application appointment, when their examination was completed at a previous date (within 6 months).

Inclusion Criteria:

* American Society of Anesthesiologist (ASA) Classification I or II
* Ages 5 to 14 years
* Cooperative behavior at present visit or recorded at the previous encounter (classified as 3 or 4 on the Frankl Behavioral Rating Scale).
* At least one erupted caries-free permanent molar in each quadrant
* Ability able to speak and understand English or Spanish
* There will be no exclusions based on race, gender, and ethnicity.

Exclusion Criteria:

* ASA Classification III or higher
* Uncooperative behavior at present visit or recorded at the previous encounter (classified as 1 or 2 on the Frankl Behavioral Rating Scale).
* Patients who require less than four sealants on permanent molars
* Patients who do not provide assent or consent.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nuntiya Kakanantadilok, DMD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collette J, Wilson S, Sullivan D. A study of the Isolite system during sealant placement: efficacy and patient acceptance. Pediatr Dent. 2010 Mar-Apr;32(2):146-50. PMID 20483019
- [Background] Alhareky MS, Mermelstein D, Finkelman M, Alhumaid J, Loo C. Efficiency and patient satisfaction with the Isolite system versus rubber dam for sealant placement in pediatric patients. Pediatr Dent. 2014 Sep-Oct;36(5):400-4. PMID 25303507
- [Background] Beauchamp J, Caufield PW, Crall JJ, Donly K, Feigal R, Gooch B, Ismail A, Kohn W, Siegal M, Simonsen R; American Dental Association Council on Scientific Affairs. Evidence-based clinical recommendations for the use of pit-and-fissure sealants: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2008 Mar;139(3):257-68. doi: 10.14219/jada.archive.2008.0155. PMID 18310730
- [Background] Lyman T, Viswanathan K, McWhorter A. Isolite vs cotton roll isolation in the placement of dental sealants. Pediatr Dent. 2013 May-Jun;35(3):E95-9. PMID 23756302
- [Background] Primosch RE, Barr ES. Sealant use and placement techniques among pediatric dentists. J Am Dent Assoc. 2001 Oct;132(10):1442-51; quiz 1461. doi: 10.14219/jada.archive.2001.0061. PMID 11680361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were selected from pediatric patients who presented to one of the four Montefiore pediatric dental clinics for an intake or a recall visit and who were determined to benefit from sealants application, or from patients who present solely for a sealant application appointment, when their examination was done at a previous date (within 6 months).
Groups:
- Cotton Roll Isolation (Left) First, Then Dryshield Isolation (Right): Group (1) Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using Dryshield (DS) on the right side.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
  The four arms/groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Cotton Roll Isolation (Right) First, Then Dryshield Isolation (Left): Group (2) Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using Dryshield (DS) on the left side.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Dryshield Isolation (Left) First, Then Cotton Roll Isolation (Right): Group (3) Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using cotton rolls (CRI) on the right side.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Dryshield Isolation (Right) First, Then Cotton Roll Isolation (Left): Group (4) Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using cotton rolls (CRI) on the left side.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
Period: Overall Study
Arm/Group | Cotton Roll Isolation (Left) First, Then Dryshield Isolation (Right) | Cotton Roll Isolation (Right) First, Then Dryshield Isolation (Left) | Dryshield Isolation (Left) First, Then Cotton Roll Isolation (Right) | Dryshield Isolation (Right) First, Then Cotton Roll Isolation (Left)
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cotton Roll Isolation (Left) First, Then Dryshield Isolation (Right): Group (1) Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using Dryshield (DS) on the right side.
  The four arms/groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Cotton Roll Isolation (Right) First, Then Dryshield Isolation (Left): Group (2) Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using Dryshield (DS) on the left side.
  The four arms/groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Dryshield Isolation (Left) First, Then Cotton Roll Isolation (Right): Group (3) Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using cotton rolls (CRI) on the right side.
  The four arms/groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Dyshield Isolation (Right) First, Then Cotton Roll Isolation (Left): Group (4) Dryshield (DS) was be used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using cotton rolls (CRI) on the left side.
  The four arms/groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Total: Total of all reporting groups
Arm/Group | Cotton Roll Isolation (Left) First, Then Dryshield Isolation (Right) | Cotton Roll Isolation (Right) First, Then Dryshield Isolation (Left) | Dryshield Isolation (Left) First, Then Cotton Roll Isolation (Right) | Dyshield Isolation (Right) First, Then Cotton Roll Isolation (Left) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Full Range); unit: years] | 8.6 [7 to 10] | 8.6 [6 to 11] | 8.8 [6 to 13] | 8.5 [6 to 12] | 8.6 [6 to 13]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Forms used to extract study-related data from patient files did not capture gender/sex. The forms were de-identified so it was not possible to track back to the original patient records to retrieve gender/sex data.
  Participants
    Unknown | 8 | 8 | 8 | 8 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Placement Time of Sealants Using Dryshield (DS) vs Cotton Rolls (CRI)
Description: The time for sealant application was recorded with a stopwatch by the dental assistant as follows for the techniques: the insertion of the first isolation aid (CRI or DS) in the oral cavity constituted the start time, and the end time was when the corresponding isolation aid (CRI or DS) was removed from the oral cavity after the sealants application.
Time Frame: Initial insertion of isolation aid (CRI or DS) and removal of corresponding isolation aid (CRI or DS)
Population: Results were analyzed and reported based on the sequence the interventions were administered.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Cotton Roll Isolation (Left): Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using Dryshield (DS) on the opposite side.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
- Cotton Roll Isolation (Right): Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using Dryshield (DS) on the opposite side.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
- Dryshield Isolation (Left): Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
- Dryshield Isolation (Right): Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
Arm/Group | Cotton Roll Isolation (Left) | Cotton Roll Isolation (Right) | Dryshield Isolation (Left) | Dryshield Isolation (Right)
Number analyzed (Participants) | 16 | 16 | 16 | 16
Seconds | 164.88 (28.78) | 160.50 (26.00) | 164.56 (27.72) | 167.81 (28.92)

2. Primary Outcome: Patient Preference as Assessed by Verbal Self-report Survey
Description: Right after the procedure, participants completed a verbal survey. The survey consisted of seven closed-ended questions intended to assess the participants' opinion on things such as comfort, noise, taste, and tissue stretching. Some survey questions require a YES or NO answer (i.e. Did you taste any of the materials used?). Other questions required the participant to select CRI or DS (i.e. Which system was the most comfortable?). The pediatric dental attending asked each patient each question, in the same sequence.
  Patient preferences were assessed with Question number 4, which specifically asked " If we did the procedure again, which system would you prefer?" The options were the Cotton Roll Isolation (CRI) or the Dryshield (DS) system. The reported values represents the response to Question number 4.
Time Frame: Immediately after the dental procedure is completed, up to 30 minutes
Population: All 32 participants who were enrolled into the study were queried for their preference (CRI vs DS). Only 8 participants per group analyzed (instead of 16 as in the other Primary Outcome Measure) as the survey was only administered once per participant.
Measure: Count of Participants; unit: Participants
Groups:
- Cotton Roll Isolation (Left) First, Then Dryshield Isolation (Right): Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using Dryshield (DS) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Cotton Roll Isolation (Right) First, Then Dryshield Isolation (Left): Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using Dryshield (DS) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Dryshield Isolation (Left) First, Then Cotton Roll Isolation (Right): Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the left side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
- Dryshield Isolation (Right) First, Then Cotton Roll Isolation (Left): Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  The four groups are a result of randomizing the side receiving one of the interventions (CRI v. DS) as well as the order of application (first v. second) resulting in a 1:1:1:1 randomization ratio with each patient acting as their own control.
Arm/Group | Cotton Roll Isolation (Left) First, Then Dryshield Isolation (Right) | Cotton Roll Isolation (Right) First, Then Dryshield Isolation (Left) | Dryshield Isolation (Left) First, Then Cotton Roll Isolation (Right) | Dryshield Isolation (Right) First, Then Cotton Roll Isolation (Left)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  Cotton Roll Isolation (CRI) | 7 | 4 | 5 | 1
  Dryshield (DS) | 1 | 4 | 3 | 7

ADVERSE EVENTS:
Time Frame: During Dental sealant appointment (average about 30 minutes)
Description: Adverse events were summarized/categorized for the four Arms/Groups based on the sequence the interventions were placed.
Groups:
- Cotton Roll Isolation (Right): Cotton rolls (CRI) were used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using Dryshield (DS) on the opposite side.
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water is used.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time.
- Dryshield Isolation (Right): Dryshield (DS) was used to isolate the maxillary and mandibular teeth on the right side of the mouth, followed by sealants placement using cotton rolls (CRI) on the opposite side.
  Dryshield: DryShield (DS) is an all-in-one isolation system. It combines the tasks of fluid evacuation, tongue and cheek retraction, and serves as a bite block. Its design allows it to suction and isolate half the oral cavity at a time
  Cotton rolls: Cotton Roll Isolation requires placing cotton rolls along the buccal mucosa, especially over the parotid glands ducts for maxillary teeth. For the mandibular teeth, the cotton rolls are placed in the buccal vestibule and the floor of the mouth (between the lower buccal mucosa and underneath and/or between the tongue). With this technique, a high-speed evacuation of saliva and water was used.
Arm/Group | Cotton Roll Isolation (Left) | Cotton Roll Isolation (Right) | Dryshield Isolation (Left) | Dryshield Isolation (Right)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT02995369/Prot_SAP_000.pdf